CLINICAL TRIAL: NCT06192199
Title: The Diagnostic Value of APTT/Fibrinogen Ratio in Pulmonary Embolism
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-501
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-01

CONDITIONS: Acute Pulmonary Embolism
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute pulmonary embolism
  Interventions: Diagnostic Test: 2018 edition of the Guidelines for Diagnosis
- Patients without acute pulmonary embolism
  Interventions: Diagnostic Test: 2018 edition of the Guidelines for Diagnosis

INTERVENTIONS:
Diagnostic Test: 2018 edition of the Guidelines for Diagnosis — According to the 2018 edition of the Guidelines for Diagnosis, Treatment and Prevention of Pulmonary Thromboembolism, and based on inclusion and exclusion criteria, enrolled patients were divided into a pulmonary embolism group and a non pulmonary embolism group

SUMMARY:
From January 1, 2023 to December 30, 2023, patients who were suspected of pulmonary embolism and underwent CTPA examination at Nanyang Hospital of Southern Medical University were divided into pulmonary embolism group and non pulmonary embolism group. 1. Collect relevant data, including gender, age, primary disease, CTPA imaging and reports, BNP, troponin, electrocardiogram, cardiac ultrasound, PT, APTT, TT, fibrinogen, D-dimer, etc., and analyze demographic data, pulmonary embolism risk grading, APTT/fibrinogen ratio, and determine their cut-off values through statistical analysis of the two groups. 2. Follow up on the APTT/fibrinogen ratio after anticoagulation treatment and bleeding in the pulmonary embolism group.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent form;
2. When signing the informed consent form, the age is equal to or greater than 18 years old, regardless of gender;
3. From January 1, 2023 to December 30, 2023, the patient was diagnosed with suspected pulmonary embolism at the Southern Hospital of Southern Medical University and underwent enhanced pulmonary artery scanning examination.

Exclusion Criteria:

1. Patients with gastrointestinal bleeding, severe trauma, acute coronary syndrome, severe liver disease (childC grade), and coagulation dysfunction;
2. Patients with pulmonary embolism diagnosed outside the hospital and regular anticoagulation;
3. Patients undergoing regular anticoagulant therapy such as atrial fibrillation and valve replacement;
4. Patients deemed unsuitable for participation in this study by the researchers.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From January 1, 2023 to December 30, 2023, the patients were diagnosed with suspected pulmonary embolism at the Southern Hospital of Southern Medical University and underwent enhanced pulmonary artery scanning examination. According to the 2018 edition of the Guidelines for Diagnosis, Treatment and Prevention of Pulmonary Thromboembolism, and based on inclusion and exclusion criteria, enrolled patients were divided into a pulmonary embolism group and a non pulmonary embolism group
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cutoff value of APTT/FIB between patients with and without acute pulmonary embolism | 2024.01-2026.12

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital of Southern Medical University, Guangzhou, Guangdong, China